CLINICAL TRIAL: NCT00248391
Title: The Influence of Feeding Position on Pulmonary Morbidity in Young Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None
Other Study IDs: avitalbotlitis- HMO-CTIL; no grant meanwhile
Record Dates: First submitted 2005-11-03; First posted 2005-11-04 (Estimated); Last update posted 2007-10-26 (Estimated); Status verified 2006-10

CONDITIONS: Pulmonary Diseases; Tonsillar Hypertrophy; Otitis Media; Dental Caries
Keywords: adenoid hypertrophy; feeding position; supine; upright; pneumonia; wheezing; otitis; adenoid; tonsil; caries
MeSH Terms: conditions — Lung Diseases; Otitis Media; Dental Caries; Deception; Pneumonia; Respiratory Sounds; Otitis

INTERVENTIONS:
Behavioral: upright feeding

SUMMARY:
Supine feeding position is associated with serous otitis media. The hypothesis is that supine feeding is associated with recurrent otitis media, tonsillar and adenoid hypertrophy and recurrent pneumonia secondary to recurrent aspiration.

DETAILED DESCRIPTION:
The aim of the study is to compare two "mother and child health clinic" stations with similar socioeconomic background. Mothers from the study station will be instructed to feed their children only in an upright position since birth. In the control station mothers will continue to feed their children as usual. Pulmonary morbidity will be evaluated prospectively through the computer system of the insurance companies.

ELIGIBILITY:
Inclusion Criteria:

* Newborn
* Mother's compliance

Exclusion Criteria:

* Bronchopulmonary dysplasia (BPD)
* Asthma
* Cystic fibrosis
* Heart disease

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2000 (Estimated)
Dates: Study Completion 2008-01 (Estimated)

PRIMARY OUTCOMES:
pulmonary and ear-throat-nose morbidity
medical costs | measured every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Avraham Avital, Prof, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel